CLINICAL TRIAL: NCT01351506
Title: Effect and Determinant Level of Admission Body Weight and Daily Weight Change and Prognoses of Critically and High Risk Surgical Patients
Brief Title: Effect of Body Weight Change to Surgical ICU Outcomes
Status: Completed | Type: Observational
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kaweesak Chittawatanarat, Department of Surgery, Chiang Mai University
Other Study IDs: 10FEB010924
Record Dates: First submitted 2011-05-09; First posted 2011-05-11 (Estimated); Results first posted 2014-11-07 (Estimated); Last update posted 2014-11-07 (Estimated); Status verified 2014-11

CONDITIONS: Body Weight; Weight Change
Keywords: Body weight; Body mass index; Weight change; ICU outcomes
MeSH Terms: conditions — Body Weight; Body Weight Changes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Aims of study

1. Effect of daily weight change upto 7 days from ICU admission to outcome of treatment in 28 days
2. Determination cut point of maximum weight change to outcome treatment

DETAILED DESCRIPTION:
Study type : Prospective observational study Location : General surgical intensive care unit Inclusion criteria : All admission patient with expected survive more than 24 hours Exclusion criteria : Patient died within 24 hours or who could not be weighed.

ELIGIBILITY:
Inclusion Criteria:

* All admitted ICU patients expected survive more than 24 hours

Exclusion Criteria:

* All expected ICU patients survive less than 24 hours
* All patient cannot be weighed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All admitted ICU patients which expected survive more than 24 hours.
Sampling Method: Non-Probability Sample
Enrollment: 465 (Actual)
Dates: Start 2011-05; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kaweesak Chittawatanarat Assistant Professor, Principal Investigator — Chaing Mai University
Locations (1):
- Department of Surgery, Faculty of Medicine, Maharaj Nakorn Chiang Mai hospital, Muang Chiang Mai, Chiang Mai, Thailand

REFERENCES:
- [Derived] Chittawatanarat K, Pichaiya T, Chandacham K, Jirapongchareonlap T, Chotirosniramit N. Fluid accumulation threshold measured by acute body weight change after admission in general surgical intensive care units: how much should be concerning? Ther Clin Risk Manag. 2015 Jul 27;11:1097-106. doi: 10.2147/TCRM.S86409. eCollection 2015. PMID 26251605

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort Patient: A total of 602 patients as inclusion criteria between May 2011 and August 2012 were enrolled on the ICU admission (day 0). One hundred thirty seven patients were excluded due to a short stay in ICU or were not weighed a second time on day 1. The remainder of 465 patients were included and followed in this study.
Period: Overall Study
Arm/Group | Cohort Patient
Started | 602
Completed | 465
Not Completed | 137

BASELINE CHARACTERISTICS:
Groups:
- ICU Survivors: Patients who survivors from ICU discharge status
- ICU Non Survivors: Patients who non survivors from ICU discharge status
- Total: Total of all reporting groups
Arm/Group | ICU Survivors | ICU Non Survivors | Total
Number analyzed (Participants) | 395 | 70 | 465
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60 [49 to 72] | 53 [45 to 74] | 60 [49 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 148 | 31 | 179
  Male | 247 | 39 | 286

OUTCOME MEASURES:

1. Primary Outcome: In Hospital Mortality
Description: 28 days mortality if patient still have be admitted in hospital.
Time Frame: within 28 days after ICU admission to dead
Population: Total 465 patients
Measure: Number; unit: participants
Groups:
- </= 5%: Maximum weight change upto 7 days less than or equal to 5% of admission body weight
- > 5%: Maximum weight change upto 7 days more than 5% of admission weight
Arm/Group | </= 5% | > 5%
Number analyzed (Participants) | 306 | 159
participants | 52 | 44

2. Secondary Outcome: Re Intubation Within 72 Hours
Description: Patient who need re-intubation within 72 hours
Time Frame: ICU complications up to 28 days after ICU admission
Population: All
Measure: Number; unit: participants
Arm/Group | </= 5% | > 5%
Number analyzed (Participants) | 306 | 159
participants | 12 | 15

3. Secondary Outcome: Acute Kidney Injury
Description: New acute kidney injury in ICU
Time Frame: Acute kidney injury
Measure: Number; unit: participants
Arm/Group | </= 5% | > 5%
Number analyzed (Participants) | 306 | 159
participants | 68 | 51

ADVERSE EVENTS:
Time Frame: up to 28 days after ICU admission
Description: Events occurring within 28 days after ICU admission
Arm/Group | </= 5% | > 5%
Serious Adverse Events (participants affected / at risk) | 11/306 | 19/159
Other Adverse Events (participants affected / at risk) | 38/306 | 37/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | </= 5% (N=306) | > 5% (N=159)
Renal replacement therapy (Renal and urinary disorders) | 11 (11) | 19 (19) — Require of renal replacement therapy
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | </= 5% (N=306) | > 5% (N=159)
Delirium (Nervous system disorders) | 38 (38) | 37 (37) — Delirium at least 4 of following criteria: 1) consciousness alteration, 2) inattention, 3) disorientation, 4) hallucination- delusion- psychosis, 5) psychomotor agitation or retardation, 6) inappropriate speech or mood, and 7) symptom fluctuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes